CLINICAL TRIAL: NCT00007332
Title: A Phase II Clinical Trial to Evaluate the Immunogenicity and Safety of a Combined Regimen Using ALVAC vCP1452 and AIDSVAX B/B
Brief Title: Safety and Immune Response Study of the Vaccine ALVAC vCP1452 Alone or in Combination With AIDSVAX B/B
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: Double | Purpose: Prevention
Other Study IDs: HVTN 203; AVEG 203; 10596 (Registry Identifier: DAIDS ES Registry Number); NCT00006147 (obsolete NCT alias)
Record Dates: First submitted 2000-12-16; First posted 2001-08-31 (Estimated); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; HIV Envelope Protein gp120; AIDS Vaccines; CD8-Positive T-Lymphocytes; HIV Seronegativity; AIDSVAX; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Biological: ALVAC(2)120(B,MN)GNP (vCP1452)
Biological: MN rgp120/HIV-1 and GNE8 rgp120/HIV-1

SUMMARY:
The purpose of this study is to see if the vaccines tested are safe when given alone and when given together, and how the immune system responds to the vaccines.

Vaccines are given to people to try to prevent an infection or disease. Early testing in a few people has shown that the HIV vaccines ALVAC vCP1452 and AIDSVAX B/B seem to be safe to use.

DETAILED DESCRIPTION:
There is no cure for HIV infection or AIDS, and drug therapy is too expensive for most affected populations. For this reason, the development of safe, effective vaccines to prevent HIV infections worldwide is needed. ALVAC vCP1452 and MN rgp120/HIV-1 have been shown to be well tolerated in Phase I and II studies. ALVAC vCP1452 given alone or in combination with subunit antigens [AS PER AMENDMENT 10/12/00: antigen] is a candidate vaccine to be evaluated for the ability to produce and express vaccine antigen in greater quantity for a longer time and with improved immunogenicity.

Volunteers are randomized to 1 of 7 [AS PER AMENDMENT 10/12/00: 1 of 4] groups and stratified by risk status. Prior to immunization, evaluations and blood draws are done to monitor hematological, chemical, and immunologic parameters. Volunteers receive 2 injections of the following vaccines at Months 0, 1, 3, and 6:

Group A: ALVAC vCP1452 and alum placebo [AS PER AMENDMENT 10/12/00: AIDSVAX placebo (aluminum hydroxide adjuvant)] at Months 0, 1, 3, and 6.

Group B: ALVAC vCP1452 and alum placebo [AS PER AMENDMENT 10/12/00: AIDSVAX placebo] at Months 0 and 1 and ALVAC vCP1452 and AIDSVAX B/B at Months 3 and 6.

Group C: ALVAC placebo and alum placebo. [AS PER AMENDMENT 10/12/00: ALVAC vCP1452 and AIDSVAX B/B at Months 0, 1, and 6 and ALVAC vCP1452 and AIDSVAX placebo at Month 3.] Group D: ALVAC vCP1452 and alum placebo at Months 0 and 1 and ALVAC vCP1452 and MN rgp120 at Months 3 and 6. [AS PER AMENDMENT 10/12/00: ALVAC placebo and AIDSVAX placebo at Months 0, 1, 3, and 6.] Group E: ALVAC vCP1452 and AIDSVAX B/B at Months 0, 1, and 6; ALVAC vCP1452 and alum placebo at Month 3. [AS PER AMENDMENT 10/12/00: Group E has been discontinued.] Group F: ALVAC vCP1452 and AIDSVAX B/B. [AS PER AMENDMENT 10/12/00: Group F has been discontinued.] Group G: ALVAC vCP1452 and alum placebo at Months 0 and 1; ALVAC vCP1452 and AIDSVAX B/E at Months 3 and 6. [AS PER AMENDMENT 10/12/00: Group G has been discontinued.] Following each pair of injections, volunteers are observed in the clinic for 30 minutes. Volunteers keep a record of body temperature and any other symptoms and report results to their AIDS Vaccine Evaluation Unit. Evaluations are performed by telephone or clinic visit on Days 1 and 2 after each vaccination. [AS PER AMENDMENT 10/12/00: Volunteers record all relevant signs and symptoms occurring 48 hours after each vaccination and provide that information at each clinic visit.] HIV testing is conducted every 3 to 6 months and volunteers are asked to complete social harms questionnaires once at Day 168 and once at the end of the study. Volunteers are followed on the study for a minimum of 18 months after the first immunization. Safety is evaluated by closely monitoring for local and systemic adverse reactions during the course of the trial.

ELIGIBILITY:
Inclusion Criteria

Volunteers may be eligible for this study if they:

* Are HIV-negative.
* Are 18 to 60 years old.
* Have a CD4 cell count of 400 cells/mm3 or more.
* Agree to use adequate birth control for 1 month before study entry and during the study (female participants).
* Have a normal history and physical examination.
* Are available for 12 months of follow-up for the planned duration of the study.
* Have a negative pregnancy test within 3 days prior to injections.

Exclusion Criteria

Volunteers will not be eligible for this study if they:

* Are pregnant or breast-feeding.
* Have chronic hepatitis B.
* Are taking medications that affect the immune system.
* Have an immune system problem, any long-term illness, or any autoimmune disease.
* Have cancer, except if it has been removed with surgery and cure is likely.
* Have a physical condition, mental condition, or job or work that may interfere with the study.
* Have been suicidal, or have ever needed medicines for a serious mental condition.
* Have received certain vaccines within 60 days of study entry.
* Have used experimental drugs within 30 days prior to study entry.
* Have received any blood products, such as immunoglobulin, in the last 6 months.
* Have active syphilis.
* Have active tuberculosis.
* Have history of severe allergy or any serious reactions to vaccines.
* Have had HIV-1 vaccines in a clinical study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 330
Dates: Study Completion 2003-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barney Graham, Study Chair
Locations (17):
- United States (17):
  - Alabama Vaccine CRS, Birmingham, Alabama
  - San Francisco Dept. of Public Health, San Francisco Gen. Hosp., San Francisco, California
  - San Francisco Vaccine and Prevention CRS, San Francisco, California
  - Project Brave HIV Vaccine CRS, Baltimore, Maryland
  - Johns Hopkins Bloomberg School of Public Health, Ctr. for Immunization Research, Project SAVE-DC, Baltimore, Maryland
  - Johns Hopkins Bloomberg School of Public Health,Ctr for Immunization Research,Project SAVE-Baltimore, Baltimore, Maryland
  - Brigham and Women's Hosp. CRS, Boston, Massachusetts
  - Fenway Community Health Clinical Research Site (FCHCRS), Boston, Massachusetts
  - Saint Louis Univ. School of Medicine, HVTU, St Louis, Missouri
  - HIV Prevention & Treatment CRS, New York, New York
  - NY Blood Ctr./Union Square CRS, New York, New York
  - Univ. of Rochester HVTN CRS, Rochester, New York
  - NY Blood Ctr./Bronx CRS, The Bronx, New York
  - Miriam Hospital's HVTU, Providence, Rhode Island
  - Vanderbilt Vaccine CRS, Nashville, Tennessee
  - Infectious Diseases Physicians, Inc., Annandale, Virginia
  - FHCRC/UW Vaccine CRS, Seattle, Washington